CLINICAL TRIAL: NCT06443138
Title: Preparation for Medical and Surgical Procedures in Oncogeriatry. Pilote Study PRIMECHO
Brief Title: Preparation for Medical and Surgical Procedures in Oncogeriatry.
Acronym: PRIMECHO
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 23-AOIP-03
Record Dates: First submitted 2024-05-23; First posted 2024-06-05 (Actual); Last update posted 2024-12-09 (Actual); Status verified 2024-12

CONDITIONS: Geriatric Oncology
Keywords: ederly; cancer
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Intervention Model Description: Implementation of a personalized pre-habilitation program at home before surgery
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Personalized pre-habilitation program (Experimental)
  Interventions: Other: Personalized pre-habilitation program

INTERVENTIONS:
Other: Personalized pre-habilitation program — Each patient will undergo 4 weeks of individualized pre-habilitation before surgery.
  Each session (1 session per day) will be carried out autonomously by the patient at home, via a dedicated application (Activiti Pro) installed on their tablet or smartphone.

SUMMARY:
Surgical management is one of the most frequently used interventions in the treatment of many cancers, but it can be associated with a high risk of postoperative complications.

The maintenance and optimization of functional abilities before, during and after treatment are major for elderly cancer patients, as it is now well established that there is a link between the level of functional capacity and the occurrence of these complications.

The scientific literature shows that the benefits of pre- and post-operative training programs, but these benefits only apply to a fraction of the patients adhering to the programs. The modalities of intervention (training load, follow-up, etc.) as well as patient involvement in these programs are major issues that need to be addressed to optimize their benefits.

Individualizing pre-habilitation, on the basis of the management of the training load, and therefore objective fatigue, would enable better patient adherence to the program, and optimize its benefits.

In this context, the PRIMECHO project aims to individualize pre-habilitation in order to improve functional of patients in the pre-habilitation or accelerated recovery after surgery phase. The aim is for the patient to be in optimum physical condition at the time of the intervention or treatment.

ELIGIBILITY:
Inclusion Criteria:

* Patient aged 70 or over
* Cancer patient with planned surgery,
* Mini Mental State Examination score greater than or equal to 24 (performed in advance by the geriatrician),
* Patient affiliated to or benefiting from a social security insurance
* Signed free and informed consent.

Exclusion Criteria:

* Inability to walk or perform unsupervised exercises.
* Vulnerable people

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-11-06 (Actual); Primary Completion 2026-11-10 (Estimated); Study Completion 2026-11-10 (Estimated)

PRIMARY OUTCOMES:
Maximal walking distance to 6 -MWT | at inclusion
  Metres walked during 6 minutes
Maximal walking distance to 6 -MWT | at 4 weeks
  Metres walked during the test
Maximal walking distance to 6 -MWT | at 8 weeks
  Metres walked during the test
Maximal walking distance to 6 -MWT | at 16 weeks
  Metres walked during the test

SECONDARY OUTCOMES:
EORTC-QLQC30 | at inclusion, 4 weeks, 8 weeks, 16 weeks
  QLQC30 is a 30-item instrument designed to measure quality of life in all cancer patients.
  It contains 30 questions and assesses the quality of life of oncological patients multidimensionally over 10 subscales. All sub-scales and the 6 individual items have a score range from 0 to 100 points. A higher score represents better function and a higher quality of life. In the symptom subscale, however, a higher score represents a higher level of symptoms or problems. Since there is no total score, all subscales and the individual items must be considered individually and evaluated using normative data.
Fatigue scale (MFI-20) | at inclusion, 4 weeks, 8 weeks, 16 weeks
  Multidiensional Fatigue Inventory-20 (MFI-20) questionnaire. 5 scales. Higher scores means worse outcome.
  General Fatigue dimension: Minimum value: 4. Maximum Value: 20. Physical fatigue dimension: Minimum value: 4. Maximum Value: 20. Reduced activity dimension: Minimum value: 4. Maximum Value: 20. Reduced motivation dimension: Minimum value: 4. Maximum Value: 20. Mental fatigue dimension: Minimum value: 4. Maximum Value: 20.
Internationnal Physiqual activity questionaire (IPAQ-short) | at inclusion, 4 weeks, 8 weeks, 16 weeks
  This questionnaire assesses overall physical activity and sedentary time over the last seven days. The questionnaire looks at intense, moderate and walking activity, as well as time spent sitting down (sedentary lifestyle), whether during leisure activities, at work, in daily life or during transport.
  The questionnaire composed with 7 questions classifies the subject according to 3 levels of activity: inactive, moderate, high.

CONTACTS AND LOCATIONS:
Overall Officials: Rabia Boulahssass, MD, Principal Investigator — Centre Hospitalier Universitaire de Nice
Locations (1):
- CHU de Nice, Nice, France

IPD SHARING:
Plan to Share IPD: Undecided